CLINICAL TRIAL: NCT04135404
Title: Factors That Impact the Relationship Between Pulmonary Status and Actual Electronic Cigarette Use (Secondary Data Analysis)
Brief Title: Factors That Impact the Relationship Between Pulmonary Status and Actual Electronic Cigarette Use
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mohammed Alqahtani, Ph.D. Candidate, Rehabilitation Science Program, University of Alabama at Birmingham
Other Study IDs: IRB 300003376
Record Dates: First submitted 2019-10-18; First posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Electronic Cigarette Use; Pulmonary Disease
MeSH Terms: conditions — Vaping; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pulmonary Group: This project will be achieved by using a publicly available data set (Behavioral Risk Factor Surveillance System, 2017). The subjects from the data set will be selected on their pulmonary status; pulmonary group are those who have reported any pulmonary diseases and they will be included in this study as pulmonary group.
  Interventions: Other: health-related telephone surveys
- Control Group: This project will be achieved by using a publicly available data set (Behavioral Risk Factor Surveillance System, 2017). The subjects from the data set will be selected on their pulmonary status; The control group are subjects without pulmonary diseases and they will be included as (control group).
  Interventions: Other: health-related telephone surveys

INTERVENTIONS:
Other: health-related telephone surveys — The Behavioral Risk Factor Surveillance System (BRFSS) is a health-related telephone surveys that collect state data about United States residents regarding their health-related risk behaviors, chronic health conditions, and use of preventive services (Secondary-data analysis).

SUMMARY:
Secondary data analysis will be performed as our approach to complete the study. A nationally representative dataset (BRFSS, 2017) will be used to answer the above hypotheses.

DETAILED DESCRIPTION:
Secondary data analysis will be performed as our approach to complete the study. A nationally representative dataset (BRFSS, 2017) will be used to answer our research questions. Our rationale is that there is insufficient research assessing the relationship between pulmonary status and e-cigarette use and that some factors, such as behavioral variables or psychosocial variables, might influence this relationship. Our expectation is that this study will deepen the understanding of the relationship between pulmonary status and e-cigarette use among U.S. adults. This study will cast light on different factors that influence the relationship between pulmonary status and e-cigarette use. Also, the following secondary outcomes will be tested: Severity of COPD symptoms (COPD group) moderate the relationship between pulmonary status (COPD status) and e-cigarette use, and Severity of asthma symptoms (asthma group) moderate the relationship between pulmonary status (asthma status) and e-cigarette use.

ELIGIBILITY:
This is secondary data analysis, so there is no control over the data (inclusion criteria, and exclusion criteria).

Inclusion Criteria:

Group 1: Pulmonary

* Are 18 years of age or older.
* Reported any of the pulmonary disease (Asthma, COPD). Group 2: Control Group
* Are 18 years of age or older.
* Free from any pulmonary disease (asthma, COPD).

Exclusion Criteria Group 1: Pulmonary

* Are younger than 18 years of age.
* Did not report any of the pulmonary disease (Asthma, COPD). Group 2: Control Group
* Are younger than 18 years of age.
* Reported any pulmonary disease (asthma, COPD

The Behavioral Risk Factor Surveillance System (BRFSS) is health-related telephone surveys that collect state data about United States residents regarding their health-related risk behaviors, chronic health conditions, and use of preventive services. This database contains data to help determine e-cigarette use in individuals with pulmonary disease in the US which little is known.

Note: The Behavioral Risk Factor Surveillance System (BRFSS) is a public dataset, and the data is publicly available online at (https://www.cdc.gov/brfss/annual_data/annual_2017.html)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * This study will use a quantitative, cross-sectional research design. The project has two phases for completion.
  * This project will be achieved by using a publicly available dataset (Behavioral Risk Factor Surveillance System, 2017). The subjects from the dataset will be selected on their pulmonary status; subjects without pulmonary diseases and those who have reported any pulmonary diseases will be included in this study
Sampling Method: Probability Sample
Enrollment: 400000 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Poor mental health mediate the relationship between pulmonary status (pulmonary vs. non-pulmonary) and e-cigarette use. | 1 year
  This question assesses mental health, including stress, depression, and emotional problems, by asking participants the number of days out of the last 30 days that their mental health was not good (continuous variables).
Smoking mediate the relationship between pulmonary status (pulmonary vs. non-pulmonary) and e-cigarette use. | 1 year
  Smoking: This scale assesses the frequency of smoking cigarettes: 1 = every day, 2 = some days, 3 = not at all.
E-cigarette use (Dependent Variable) | 1 year
  This survey item asks participants if they ever used an e-cigarette or other electronic "vaping" product, even just one time, in their entire life (Yes/No).
Alcohol use moderate the relationship between pulmonary status (pulmonary vs. healthy) and e-cigarette use | 1 year
  This question assesses the number of days in the last 30 days that participants have drunk alcohol (continuous variables).
(healthy days (health-related quality of life) mediate the relationship between pulmonary status (pulmonary vs. non-pulmonary) and e-cigarette use. | 1 year
  In reference to healthy days, these questions assess health-related quality of life, which is going to be assessed by asking questions concerning the number of days out of the last 30 days that the participants were physically or mentally ill (continuous variables).

SECONDARY OUTCOMES:
Marijuana use moderate the relationship between pulmonary status (pulmonary vs. healthy) and e-cigarette use. | 1 year
  This question assesses the number of days in the last 30 days that participants have used marijuana or hashish (continuous variables).
Severity of COPD symptoms (COPD group) moderate the relationship between pulmonary status (COPD, asthma) and e-cigarette use | 1 year
  Three questions are posed to assess the severity of COPD symptoms. The responses of these questions are combined to form a composite score. The first question will assess coughing, the second question will assess phlegm production, and the third question will assess shortness of breath. Answers for each of the three questions will be in a yes/no format and will be represented on a scale of 1-3, where 1 is less severe and 3 is more severe.
asthma symptoms (asthmatic group) moderate the relationship between pulmonary status (COPD, asthma) and e-cigarette use. | 1 year
  Several questions determine the severity of asthma symptoms. The first question will assess the asthma symptoms by asking the participants the number of days they were unable to work or carry out their usual activities because of their asthma symptoms (continuous variables). The second question will assess coughing, wheezing, shortness of breath, chest tightness and phlegm production by asking participants the number of days out of the last 30 that they have any of the previous symptoms (continuous variables). The final question will symptoms of asthma make it difficult for the participants to stay asleep (continuous variables).

IPD SHARING:
Plan to Share IPD: No
This is public data set, it is already published by the CDC and any researchers can use these data.
  The Behavioral Risk Factor Surveillance System (BRFSS) is a health-related telephone surveys that collect state data about United States residents regarding their health-related risk behaviors, chronic health conditions, and use of preventive services.

REFERENCES:
- [Background] Centers for Disease Control and Prevention (CDC). Behavioral Risk Factor Surveillance System Survey Data. Atlanta, Georgia: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, [2017].
- [Background] Centers for Disease Control and Prevention (CDC). Behavioral Risk Factor Surveillance System Survey Questionnaire. Atlanta, Georgia: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention, [2017]
- [Derived] Alqahtani MM, Alanazi AM, Pavela G, Dransfield MT, Wells JM, Lein DH Jr, Hendricks PS. Binge Drinking Moderates the Association Between Chronic Lung Disease and E-Cigarette Use. Respir Care. 2021 Jun;66(6):936-942. doi: 10.4187/respcare.08559. Epub 2021 Mar 9. PMID 33688091
- See also: This a comprehensive description of this data set — https://www.cdc.gov/brfss/annual_data/annual_2017.html